CLINICAL TRIAL: NCT03440788
Title: Patient-reported and Clinical Outcomes in Adults With Relapsed or Refractory Hodgkin's Lymphoma Receiving Brentuximab Vedotin: a Multicenter, Prospective, Observational Study in a Real World Setting
Brief Title: Patient-reported and Clinical Outcomes in Adults With Relapsed or Refractory Hodgkin's Lymphoma Receiving Brentuximab Vedotin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Multinational Center for Quality of Life Research, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: IISR-2017-102112
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Relapsed or Refractory Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence; Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab vedotin (BV) will be prescribed to patients in accordance with indication for treatment as second or subsequent line therapy after failure of at least one type of first-line therapy for patients with relapsed or refractory HL who are not candidates for ASCT, or for patients with relapse after ASCT within routine hematological practice. Dose, preparation, administration etc - as in Instruction for use (Prescribing information).

SUMMARY:
The goal of this is study is focusing on assessment of patient-reported outcomes in terms of quality of life (QoL) and symptom profile as well on evaluation of clinical efficacy and safety of BV in patients with refractory/resistant HL in a real-world setting.

DETAILED DESCRIPTION:
Information on QoL in patients with refractory/relapsed HL treated with BV is quite limited till now. Moreover, PRO data in patients treated for refractory/relapsed HL with BV, including long-term effects of BV on patient's QoL in a real-world setting are lacking.

The goal of this is study is focusing on assessment of patient-reported outcomes in terms of QoL and symptom profileas well on evaluation of clinical efficacy and safety of BV in patients with refractory/resistant HL in a real-world setting.

For PROs assessment QoL and symptom data will be received from patients' reports before and at 3, 6, 9, 12 months after BV treatment start and in 3 months at follow-up (15 months after base-line). The maximum duration of PRO monitoring - 15 months. To evaluate PROs the followings tools will be used: RAND SF-36 for quality of life assessment, Edmonton Symptom Assessment System (ESAS-R) for symptom assessment and Patient Global Impression of Change (PGIC) for assessment of a patient's belief about the effect of treatment.

For evaluation of response rates, duration of response, PFS and for analysis of AEs/SAEs during BV treatment the clinical data will be collected from health records at base-line, at 3, 6, 9, 12 months after BV treatment start and at 15 months of follow-up or till the last dose of BV.

No randomization and stratification will be applied. The analysis of primary (PROs assessment) and secondary outcomes (clinical outcomes) will be provided in the total patient population (n=70) and in two subgroups. The subgroups of interest will be: patients with relapsed or refractory HL who are not candidates for ASCT with prescribed treatment with BV as ≥2nd line therapy, and patients with relapse after ASCT with prescribed treatment with BV.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed diagnosis of relapsed or refractory HL
* At least 18 years of age at time of BV treatment decision
* Patients with relapsed or refractory HL who are not candidates for ASCT with prescribed treatment with BV as ≥2nd line therapy, and patients with relapse after ASCT with prescribed treatment with BV
* Patients with given informed consent
* Patients who are capable to fill out questionnaires
* Patients with expected life duration of at least 6 months

Exclusion Criteria:

* Patients enrolled in clinical trials
* Patients with contraindications to BV in accordance with instruction for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsed or refractory HL who are not candidates for ASCT and have been prescribed to treatment with BV as ≥2nd line therapy, and patients with relapse after ASCT and have been prescribed to treatment with BV. The eligibility criteria for this study are broader than for those to be treated with BV in randomized clinical trials, so as to be reflective of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in QoL and symptom severity while treatment with BV | At 3, 6, 9 and 12 months of BV treatment and at 15 months after treatment start
  The change in QoL will be assessed as the difference in QoL scales of RAND SF-36 as compared to their baseline and the difference in proportion of patients with significant negative impact on QoL. The change in symptom severity will be assessed as the difference in the severity of each ESAS-R scale and the symptom distress score as compared with their baseline value. The proportion of patients with ≥1 point improvement on ESAS-R scale will be analyzed as well.

SECONDARY OUTCOMES:
Overall response rate | At 3, 6, 9 and 12 months of BV treatment at treatment discontinuation
  Tumor response will be assessed and derived using the RESIST criteria v. 1.0.
Progression-free survival (PFS) | 15 months
  PFS will be estimated from initiation of treatment with BV till the disease progression or death from any cause.
Adverse events (AEs)/serious AEs | At 3, 6, 9 and 12 months of BV treatment
  The analysis of safety of BV will include reporting adverse events (AEs)/serious AEs (SAEs). For adverse events assessment the NCI CTCAE v. 4.0 will be used. The incidence and severity of any AEs/SAEs will be evaluated within the study

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Chelyabinsk Regional Clinical Center of Oncology and Nuclear Medicine, Chelyabinsk
  - Republican Clinical Oncology Center of the Ministry of Health of the Republic of Tatarstan, Kazan'
  - N.I. Pirogov National Medical Surgical Center, Moscow
  - Clinical Onclological Center, Omsk
  - Almazov National Medical Research Centre, Saint Petersburg
  - Raisa Gorbacheva Memorial Research Institute of Children Oncology, Hematology and Transplantation, I. P. Pavlov First Saint Petersburg State Medical University, Ministry of Health of Russia, Saint Petersburg
  - Department of occupational pathology, hematology and clinical pharmacology, V.I. Rasymovsky Saratov State Medical University, Saratov
  - Tula Regional Clinical Hospital, Tula
  - Primorskiy Regional Oncologic Center, Vladivostok